CLINICAL TRIAL: NCT00895635
Title: Exercise Training to Reduce Claudication: Arm Ergometry Versus Treadmill Walking
Brief Title: Evaluating Two Exercise Training Programs to Reduce Leg Pain in People With Peripheral Arterial Disease (The EXERT Study)
Acronym: EXERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0803M28683; R01HL090854-01A1 (NIH)
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Intermittent Claudication; Peripheral Vascular Diseases
Keywords: Claudication; Peripheral Arterial Disease; Exercise Rehabilitation; Cardiovascular Function
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treadmill Exercise Training (Experimental): Participants will take part in a 12-week supervised treadmill exercise training program.
  Interventions: Behavioral: Treadmill Exercise Training
- Arm Ergometry Exercise Training (Experimental): Participants will take part in a 12-week supervised aerobic arm ergometry exercise training program.
  Interventions: Behavioral: Arm Ergometry Exercise Training
- Usual Care Control Group (Active Comparator): Participants will receive usual care for PAD from their doctor.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Treadmill Exercise Training — 60-minute sessions of supervised treadmill exercise training three times a week for 12 weeks
  Arms: Treadmill Exercise Training
Behavioral: Arm Ergometry Exercise Training — 60-minute sessions of supervised aerobic arm exercise training using an arm ergometer three times a week for 12 weeks
  Arms: Arm Ergometry Exercise Training
Behavioral: Usual Care — Usual care for PAD
  Arms: Usual Care Control Group

SUMMARY:
Peripheral arterial disease (PAD) is a disorder that affects more than 8 million people in the United States. As a result of decreased blood flow to the legs, people with PAD may experience leg pain and difficulty with walking. This study will examine the effectiveness of two exercise programs-a treadmill walking program and an aerobic arm exercise program-at increasing walking distance and decreasing leg pain in people with PAD.

DETAILED DESCRIPTION:
PAD is a condition that occurs when atherosclerotic plaque builds up in the peripheral arteries and restricts blood flow. People with PAD often experience reduced blood flow to the legs, which may cause painful leg cramping while walking, known as intermittent claudication. Claudication affects over 4 million people in the United States, and many people with this condition can walk only ½ to 2 blocks before leg pain begins to occur. Regular treadmill walking has been shown to be effective at increasing walking distance and reducing claudication in people with PAD. However, walking on a treadmill may prove difficult for some people with PAD and usually causes increased leg pain, both of which may reduce exercise frequency. Aerobic arm exercises do not cause leg pain and may be an effective way for people with PAD to improve overall cardiovascular fitness and increase the amount of exercise they do. The purpose of this study is to compare the effectiveness of a treadmill exercise program and an aerobic arm exercise program at reducing symptoms of claudication and improving walking ability in people with PAD.

This study will enroll people with PAD and claudication. At a baseline study visit, participants will complete a treadmill walking test; a blood collection; and questionnaires to assess walking status, daily activity levels, quality of life, and mood. One week after the baseline visit, participants will attend a study visit for an assessment of forearm and leg muscle blood flow and a hand-bike test that will measure upper body strength using an arm cycle ergometer. The ergometer is a device with bicycle pedals that people move using their arms. Participants will then be randomly assigned to either a treadmill exercise training program, an arm ergometry exercise program, or a control group.

Participants in the treadmill exercise training program will attend a supervised program at one of four study sites and exercise on a treadmill for 1 hour three times a week for 12 weeks. Participants in the arm ergometry exercise program will attend a supervised program at one of four study sites and exercise using an arm cycle ergometer (hand-bike) for 1 hour three times a week for 12 weeks. Participants in both groups will also receive written instructions about exercising on their own. Participants in the control group will continue to receive usual care from their regular doctor for the treatment of PAD and will be provided with written exercise instructions. Once a week for 12 weeks, participants in the control group will attend study visits to discuss any health problems.

All participants will be asked to monitor their daily exercise for 3 separate weeks during the 12-week period by wearing an accelerometer, which will measure and record physical activity. They will also record their exercise habits in a written diary. All participants will attend study visits on 2 separate days at Weeks 6 and 12 for repeat baseline testing.

From Weeks 12 to 24, all participants will be encouraged to continue to exercise on their own at least three times a week for 30 minutes. Every 4 weeks, study researchers will call participants to offer encouragement and answer questions. At Week 23, participants will again wear an accelerometer and keep an exercise diary for 1 week. All participants will attend a final study visit at Week 24 for repeat baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Has lifestyle-limiting claudication
* Able to walk on a treadmill at 2 mph
* Able to perform arm ergometry exercise
* Able to complete a 12-week exercise program

Exclusion Criteria:

* Physical activities are limited for reasons other than claudication
* Uncontrolled high blood pressure
* Uncontrolled diabetes
* Unstable coronary heart disease
* Ischemic rest pain or tissue loss
* Recent (in the 3 months before study entry) coronary or peripheral revascularization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximal walking distance | Measured at baseline and Weeks 6, 12, and 24
Pain-free walking distance | Measured at baseline and Weeks 6, 12, and 24

SECONDARY OUTCOMES:
Limb blood flow | Measured at baseline and Weeks 6, 12, and 24
Cardiovascular function | Measured at baseline and Weeks 6, 12, and 24
Quality of life | Measured at baseline and Weeks 6, 12, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Diane J. Treat-Jacobson, PhD, RN, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States